CLINICAL TRIAL: NCT03203499
Title: A Phase 1b, Proof of Concept, Dose-Ranging Study to Evaluate the Safety of the Coadministration of Ascending Doses of ANS-6637 and Ethanol in Healthy Male Moderate Drinkers
Brief Title: A Study to Evaluate the Safety of the Coadministration of ANS-6637 and Ethanol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amygdala Neurosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANS-A-C1-001
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
Keywords: Substance abuse disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — ANS-6637

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ANS-6637 (Experimental): Single ascending doses of ANS-6637 administered orally
  Interventions: Drug: ANS-6637 Oral Tablet
- Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ANS-6637 Oral Tablet — Ascending single doses administered orally.
  Arms: ANS-6637
Drug: Placebo Oral Tablet — Placebo administered orally.
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, single-ascending-dose study to evaluate the safety and tolerability of the coadministration of up to 6 dose levels of ANS-6637 and EtOH in healthy male moderate alcohol drinkers. The study will include a screening visit, a qualification visit, a Treatment Phase and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male adults, between 21 and 45 years of age, inclusive.
2. Body mass index (BMI) within 19.0 to 34.0 kg/m2, inclusive (minimum weight of at least 50.0 kg at screening).
3. Resting semisupine vital signs at screening and each clinic admission within the following ranges:

   1. Systolic blood pressure 90 to 140 mmHg
   2. Diastolic blood pressure of 50 to 90 mmHg
   3. Heart rate of 40 to 90 beats per minute (bpm)
4. Current alcohol users who are self-reported moderate drinkers, defined as having consumed 7 to 21 standard drinks per week on average in the 6 months prior to screening and having consumed ≥5 standard drinks on at least 1 occasion in the 30 days prior to screening. One standard alcoholic drink (14 grams of EtOH) is equivalent to 43 mL (1.5 oz) hard liquor, 142 mL (5 oz) wine or 341 mL (12 oz) beer.

Exclusion Criteria:

1. Drug or alcohol dependence within the 12 months prior to screening (except nicotine), as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision (DSM-IV-TR), or any self-reported dependence or "addiction" within the subject's lifetime (except nicotine or caffeine).
2. Subjects who have ever been in treatment for substance use disorder(s) (except smoking cessation).
3. Current or prior diagnosis of any condition where alcohol consumption is contraindicated, including, but not limited to, hypertriglyceridemia, pancreatitis, liver disease, porphyria, and/or congestive heart failure, that is clinically relevant, as judged by the investigator or designee.
4. Positive urine drug test for EtOH, cocaine, oxycodone and other opioids, amphetamines, benzodiazepines and/or cannabinoids at clinic admission. Positive results may be repeated and/or subjects rescheduled at the investigator's or designee's discretion.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male moderate drinkers.
Enrollment: 48 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 36 hours postdose

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to 48 hours postdose
Time to maximum observed serum concentration (Tmax) | Up to 48 hours postdose
Areas under the plasma concentration-time curve from time zero to last quantifiable concentration (AUClast) | Up to 48 hours postdose
Ethanol Consumption | Up to 6 hours postdose
Modified 5-Item Drug Effects Questionnaire (mDEQ-5) | Up to 6 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Study Director — Vince and Associates
Locations (1):
- Vince and Associates, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No